CLINICAL TRIAL: NCT05024084
Title: Comparison of Desflurane and Sevoflurane Minimal Flow Anesthesia on Recovery Parameters and Anesthetic Depth: a Randomized Prospective Study
Brief Title: Desflurane and Sevoflurane Minimal Flow Anesthesia on Recovery and Anesthetic Depth
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Baturay Kansu Kazbek, Principal Investigator, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-009
Record Dates: First submitted 2021-08-13; First posted 2021-08-27 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Anesthesia
Keywords: general anesthesia; low flow anesthesia; sevoflurane; desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Sevoflurane (Active Comparator): The patients in this arm will be given Sevoflurane (2-3%) as volatile anesthetic throughout the duration of anesthesia.
  Interventions: Procedure: Minimal flow anesthesia (fresh gas flow <0.5 l/min) using Sevoflurane
- Group Desflurane (Active Comparator): The patients in this arm will be given Desflurane (7-8%) as volatile anesthetic throughout the duration of anesthesia.
  Interventions: Procedure: Minimal flow anesthesia (fresh gas flow <0.5 l/min) using Desflurane

INTERVENTIONS:
Procedure: Minimal flow anesthesia (fresh gas flow <0.5 l/min) using Sevoflurane — Sevoflurane will be used for the maintenance of general anesthesia which will be carried out using a fresh gas flow of less than 0,5 l/min
  Arms: Group Sevoflurane
Procedure: Minimal flow anesthesia (fresh gas flow <0.5 l/min) using Desflurane — Desflurane will be used for the maintenance of general anesthesia which will be carried out using a fresh gas flow of less than 0,5 l/min
  Arms: Group Desflurane

SUMMARY:
Minimal flow anesthesia has economic and environmental advantages in addition to providing earlier recovery following general anesthesia. There is a paucity of data concerning the effect of minimal flow anesthesia (fresh gas flow <0,5 l/min) on recovery parameters. The primary objective of this study is to compare the recovery parameters of desflurane and sevoflurane in minimal flow anesthesia while the secondary objective is to compare the effect of these agents on anesthetic depth using bispectral index.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 65
* Patients undergoing elective surgery under general anesthesia
* Patients with an American Society of Anesthesiologists Classification I or II

Exclusion Criteria:

* Patient refusal
* Emergency surgery
* Patients with a contraindication for minimal flow anesthesia
* Uncontrolled diabetes mellitus
* History of serious systemic disease (cardiac, pulmonary, hepatic)
* Utilization of another analgesic technique such as central or peripheral nerve blocks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-09-05 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Time until extubation | Up to 10 minutes after discontinuation of the volatile anesthetic
  Time interval between discontinuation of the volatile anesthetics and removal of the endotracheal tube
Time until eye opening | Up to 20 minutes after discontinuation of the volatile anesthetic
  Time interval between discontinuation of the volatile anesthetics and eye opening with verbal command
Time until transfer readiness | Up to 45 minutes after discontinuation of the volatile anesthetic
  Time interval between discontinuation of the volatile anesthetics and Aldrete score reaching 9 or greater

SECONDARY OUTCOMES:
Anesthetic depth provided by the volatile anesthetic | Change in Bispectral Index values at 5, 10, 15, 30, 60 and 120 minutes
  Anesthetic depth as measured by Bispectral Index

CONTACTS AND LOCATIONS:
Overall Officials: Baturay K Kazbek, Ass. Prof., Principal Investigator — Ufuk University Faculty of Medicine Department of Anesthesiology and Reanimation
Locations (1):
- Ufuk University Dr. Rıdvan Ege Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taskin D, Gedik E, Kayhan Z. Effects of Minimal Flow Sevoflurane or Desflurane Anaesthesia on Hemodynamic Parameters, Body Temperature and Anaesthetic Consumption. Turk J Anaesthesiol Reanim. 2020 Oct;48(5):356-363. doi: 10.5152/TJAR.2020.39699. Epub 2020 May 5. PMID 33103139
- [Background] Werner JG, Castellon-Larios K, Thongrong C, Knudsen BE, Lowery DS, Antor MA, Bergese SD. Desflurane Allows for a Faster Emergence When Compared to Sevoflurane without Affecting the Baseline Cognitive Recovery Time. Front Med (Lausanne). 2015 Oct 28;2:75. doi: 10.3389/fmed.2015.00075. eCollection 2015. PMID 26579522